CLINICAL TRIAL: NCT00745030
Title: Efficacy and Tolerability of Ramelteon in Patients With REM Behavior Disorder and Parkinsonism: A Placebo Controlled, Double Blind, Randomized, Prospective Pilot Study
Brief Title: Efficacy and Tolerability of Ramelteon in Patients With Rapid Eye Movement (REM) Behavior Disorder and Parkinsonism
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low subject recruitment and enrollment.
Sponsor: Northwestern University (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-028R
Record Dates: First submitted 2008-08-28; First posted 2008-09-01 (Estimated); Results first posted 2010-11-10 (Estimated); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: REM Behavior Disorder; Parkinsonism
Keywords: Parkinson's disease; Multiple Systems Atrophy; Lewy Body Dementia
MeSH Terms: conditions — REM Sleep Behavior Disorder; Parkinsonian Disorders; Parkinson Disease; Lewy Body Disease | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Ramelteon (TAK-375) 8mg tablets
  Interventions: Drug: Rozerem
- 2 (Placebo Comparator): Placebo 8 mg tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rozerem — Subjects take 1 8mg tablet 30 minutes before bedtime everyday for 8 weeks.
  Other Names: Ramelteon; TAK-375
  Arms: 1
Drug: Placebo — Placebo 8 mg tablets
  Arms: 2

SUMMARY:
Parkinson's disease (PD) is the second most common neurodegenerative disorder of the elderly that affects a million patients in US. Sleep dysfunction impacts up to 90% of PD patients. PD patients experience a variety of sleep disorders including parasomnias, specifically REM behavior disorder (RBD) that can precede the onset of motor manifestations of PD. RBD has negative consequences on patients' and their bed partners' quality of life mainly due to its impact on the sleep quality and day time alertness. RBD also predisposes affected individuals and their bed partners to physical injuries.

There are no FDA approved treatments for RBD. Clonazepam is the most commonly used treatment but carries risks of daytime sedation, tolerance, and withdrawal symptoms. More recently, melatonin has been demonstrated to be effective in several small studies. Ramelteon, a selective melatonin receptor agonist with favorable safety profile, could potentially be effective for the treatment of RBD.

This pilot protocol will investigate safety and efficacy of ramelteon for the treatment of RBD in subjects with parkinsonism. We plan to recruit 20 subjects with RBD diagnosed based on the clinical interview and confirmed by the polysomnographic (PSG) data. The study is designed as a prospective randomized placebo controlled 12-week study. Primary outcome measure will be change in frequency of RBD events based on the daily sleep diaries. Secondary outcome measure will be change in the amount of tonic muscle activity based on the results of the baseline and final PSG. A number of other secondary and exploratory outcome measures will be collected

DETAILED DESCRIPTION:
See above.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of parkinsonism (idiopathic PD, multiple systems atrophy, Lewy body dementia)
* RBD frequency of at least once per week based on the RBD screening clinical questionnaire
* PSG evidence of RBD
* Presence of bed partner/caregiver who sleeps in the same room as PD patient

Exclusion Criteria:

* Known hypersensitivity to ramelteon or related compounds, including melatonin and melatonin-related compounds.
* Use of hypnotics or other sedatives within a month prior to the study initiation
* Presence of active psychosis
* Use of neuroleptics, except for the atypical neuroleptics - specifically quetiapine (the dose should not exceed 50mg/day)
* Use of antidepressants unless the patient has been on a stable dose for at least three months
* Use of Venlafaxine (Effexor®)
* Presence of cognitive impairment, defined as the Mini Mental Status Examination (MMSE) score <24
* Presence of depression defined as the Beck Depression Inventory (BDI) score >14
* Significant sleep disordered breathing (defined as an apnea-hypopnea index>15 events/hr of sleep on screening PSG), significant periodic limb movement disorder (defined as a PLM index>10 events/hr of sleep with awakening on screening PSG)
* Travel through two time zones within a month prior to the study initiation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Simuni, M.D., Principal Investigator — Northwestern University, Department of Neurology; Aleksandar Videnovic, M.D., Study Director — Harvard Medical School, Associate Professor of Neurology
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Simuni T. Somnolence and other sleep disorders in Parkinson's disease: the challenge for the practicing neurologist. Neurol Clin. 2004 Oct;22(3 Suppl):S107-26. doi: 10.1016/j.ncl.2004.06.006. No abstract available. PMID 15501360
- [Background] Thorpy MJ. Sleep disorders in Parkinson's disease. Clin Cornerstone. 2004;6 Suppl 1A:S7-15. doi: 10.1016/s1098-3597(04)90013-0. PMID 15259535
- [Background] Gagnon JF, Bedard MA, Fantini ML, Petit D, Panisset M, Rompre S, Carrier J, Montplaisir J. REM sleep behavior disorder and REM sleep without atonia in Parkinson's disease. Neurology. 2002 Aug 27;59(4):585-9. doi: 10.1212/wnl.59.4.585. PMID 12196654
- [Background] Schenck CH, Bundlie SR, Patterson AL, Mahowald MW. Rapid eye movement sleep behavior disorder. A treatable parasomnia affecting older adults. JAMA. 1987 Apr 3;257(13):1786-9. PMID 3820495
- [Background] Boeve BF, Silber MH, Parisi JE, Dickson DW, Ferman TJ, Benarroch EE, Schmeichel AM, Smith GE, Petersen RC, Ahlskog JE, Matsumoto JY, Knopman DS, Schenck CH, Mahowald MW. Synucleinopathy pathology and REM sleep behavior disorder plus dementia or parkinsonism. Neurology. 2003 Jul 8;61(1):40-5. doi: 10.1212/01.wnl.0000073619.94467.b0. PMID 12847154
- [Background] Boeve BF, Silber MH, Ferman TJ, Lucas JA, Parisi JE. Association of REM sleep behavior disorder and neurodegenerative disease may reflect an underlying synucleinopathy. Mov Disord. 2001 Jul;16(4):622-30. doi: 10.1002/mds.1120. PMID 11481685
- [Background] Schenck CH, Bundlie SR, Mahowald MW. Delayed emergence of a parkinsonian disorder in 38% of 29 older men initially diagnosed with idiopathic rapid eye movement sleep behaviour disorder. Neurology. 1996 Feb;46(2):388-93. doi: 10.1212/wnl.46.2.388. PMID 8614500
- [Background] Boeve BF, Silber MH, Ferman TJ. Melatonin for treatment of REM sleep behavior disorder in neurologic disorders: results in 14 patients. Sleep Med. 2003 Jul;4(4):281-4. doi: 10.1016/s1389-9457(03)00072-8. PMID 14592300
- [Background] Takeuchi N, Uchimura N, Hashizume Y, Mukai M, Etoh Y, Yamamoto K, Kotorii T, Ohshima H, Ohshima M, Maeda H. Melatonin therapy for REM sleep behavior disorder. Psychiatry Clin Neurosci. 2001 Jun;55(3):267-9. doi: 10.1046/j.1440-1819.2001.00854.x. PMID 11422870
- [Background] Kunz D, Bes F. Melatonin as a therapy in REM sleep behavior disorder patients: an open-labeled pilot study on the possible influence of melatonin on REM-sleep regulation. Mov Disord. 1999 May;14(3):507-11. doi: 10.1002/1531-8257(199905)14:33.0.co;2-8. PMID 10348479
- [Background] Roth T, Seiden D, Sainati S, Wang-Weigand S, Zhang J, Zee P. Effects of ramelteon on patient-reported sleep latency in older adults with chronic insomnia. Sleep Med. 2006 Jun;7(4):312-8. doi: 10.1016/j.sleep.2006.01.003. Epub 2006 May 18. PMID 16709464
- [Background] Borja NL, Daniel KL. Ramelteon for the treatment of insomnia. Clin Ther. 2006 Oct;28(10):1540-55. doi: 10.1016/j.clinthera.2006.10.016. PMID 17157111
- [Background] Chaudhuri KR, Pal S, DiMarco A, Whately-Smith C, Bridgman K, Mathew R, Pezzela FR, Forbes A, Hogl B, Trenkwalder C. The Parkinson's disease sleep scale: a new instrument for assessing sleep and nocturnal disability in Parkinson's disease. J Neurol Neurosurg Psychiatry. 2002 Dec;73(6):629-35. doi: 10.1136/jnnp.73.6.629. PMID 12438461

RESULTS

PARTICIPANT FLOW:
Groups:
- Ramelteon (TAK-375) 8mg Tablets: Ramelteon (TAK-375) 8mg tablets
- Placebo 8 mg Tablets: Placebo 8 mg tablets
Period: Overall Study
Arm/Group | Ramelteon (TAK-375) 8mg Tablets | Placebo 8 mg Tablets
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ramelteon (TAK-375) 8mg Tablets | Placebo 8 mg Tablets | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (0) | 57 (7.85) | 57 (7.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in the Frequency of RBD Based on the Daily Sleep Diaries, Completed Daily for the Duration of the Study by the Study Subjects' Bed Partners/Caregivers
Description: Change in the frequency of RBD based on the daily sleep diaries, completed daily for the duration of the study by the study subjects' bed partners/caregivers.
  Data will not be analyzed. The protocol is being terminated due to low subject enrollment and recruitment.
Time Frame: 12 weeks
Population: We had difficulties with recruitment and did not manage to recruit enough participants so no data was collected and the study was terminated.
Arm/Group | Ramelteon (TAK-375) 8mg Tablets | Placebo 8 mg Tablets
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in the Amount of Tonic Muscle Activity Based on the Results of the Baseline and Final Polysomnographic (PSG) Study
Description: no participants were recruited
Time Frame: 8 weeks
Population: as for outcome 1
Arm/Group | Ramelteon (TAK-375) 8mg Tablets | Placebo 8 mg Tablets
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Ramelteon (TAK-375) 8mg Tablets | Placebo 8 mg Tablets
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No